CLINICAL TRIAL: NCT06917742
Title: A First-in-Human, Phase 1, Single-Center, Open-Label, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CPTX2309 by Intravenous Administration in Healthy Volunteers
Brief Title: A Study of CPTX2309 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Capstan Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPTX2309-01-01
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAD Cohorts (Experimental): Escalating single doses of CPTX2309 on a specified day
  Interventions: Drug: CPTX2309
- MAD Cohorts (Experimental): Escalating multiple doses of CPTX2309 on specified days
  Interventions: Drug: CPTX2309

INTERVENTIONS:
Drug: CPTX2309 — Single Escalating Dose of CPTX2309. CPTX2309 is a targeted lipid nanoparticle designed to deliver an anti-CD19 CAR mRNA preferentially to CD8+ T cells.
  Arms: SAD Cohorts
Drug: CPTX2309 — Multiple Escalating Dose of CPTX2309.CPTX2309 is a targeted lipid nanoparticle designed to deliver an anti-CD19 CAR mRNA preferentially to CD8+ T cells.
  Arms: MAD Cohorts

SUMMARY:
The purpose of this study is to assess the safety and tolerability of CPTX2309 in healthy adult participants.

DETAILED DESCRIPTION:
A first-in-human Phase 1, open label study to evaluate safety and tolerability of a single ascending dose (SAD) and multiple ascending dose (MAD) of CPTX2309 intravenously administered to healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by the investigator based on review of medical history, physical examination, and clinical laboratory tests obtained during the screening period.
* Participant is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, or clinical laboratory tests beyond what is consistent with a healthy population in the region in which the study is conducted.
* Use of any investigational medical device or investigational drug within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the first administration of CPTX2309.
* Note: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with changes in the safety parameters | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Number of participants with clinical laboratory assessment abnormalities | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Number of participants with changes in the vital signs | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Number of participants with changes in the ECG | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Number of participants who develop anti-drug antibodies (ADAs) to CPTX2309 | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Number of participants with change from baseline in vaccine antibody titers | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Changes in serum cytokine and chemokine levels that are known to be associated with CAR-T cell therapy related toxicity | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.
Change from baseline in soluble immunoglobulins (Ig) | 8 weeks
  To evaluate the safety and tolerability of CPTX2309 administered to healthy adult participants.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters | 8 weeks
  Levels of CAR+ T cells, levels of CPTX2309 components
Pharmacodynamic Parameters | 8 weeks
  Levels of circulating B cells expressed as the number of CD19 positive B cells in one microliter of blood by flow cytometry
Pharmacodynamic Parameters | 8 weeks
  Percentages of naïve and memory B cells in blood by flow cytometry
Pharmacodynamic Parameters | 8 weeks
  Levels of cytokines and chemokines in nanograms per milliliter of serum by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Farzaneh-Far, MD, Study Director — Capstan Therapeutics, Inc.
Locations (1):
- Nucleus Network Brisbane, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No